CLINICAL TRIAL: NCT06622525
Title: Use of Sodium Bicarbonate As Prophylaxis for Kidney Damage in Patients with Heatstroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General de Mexicali (Other)
Collaborators: Universidad Autonoma de Baja California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HGMexicali
Record Dates: First submitted 2024-06-06; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-06

CONDITIONS: Heat Stroke; Acute Kidney Injury; Acute Kidney Injury Due to Hypovolaemia
MeSH Terms: conditions — Heat Stroke; Acute Kidney Injury | interventions — Sodium Bicarbonate; Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized, open-label clinical trial at the General Hospital of Mexicali; central tendency measures will be obtained for variables.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): This group will receive 100 mEq of sodium bicarbonate diluted in one liter of saline solution, administered at a rate of 100 ml/h, with the goal of maintaining a urinary pH greater than 6.5.
  Interventions: Drug: Sodium bicarbonate
- Control Group (Active Comparator): This group will be manage with the usual care that is given to patients with heat stroke in this hospital.
  Interventions: Other: No intervention

INTERVENTIONS:
Drug: Sodium bicarbonate — This group will receive 100 mEq of sodium bicarbonate diluted in one liter of saline solution, administered at a rate of 100 ml/h, with the goal of maintaining a urinary pH greater than 6.5.
  Arms: Intervention Group
Other: No intervention — The usual management for heat stroke will be given to this group
  Other Names: Control Group
  Arms: Control Group

SUMMARY:
This study protocol aims to prevent the need for renal replacement therapy in patients with rhabdomyolysis secondary to heatstroke. It is based on previous studies showing that bicarbonate infusion reduces renal failure in similar contexts. The intervention will be conducted at the General Hospital of Mexicali during the summer, targeting the prevention of renal failure and reducing the necessity for renal replacement therapy.

DETAILED DESCRIPTION:
The present study protocol explores the possibility of preventing the need for renal replacement therapy in patients who develop rhabdomyolysis secondary to heatstroke. This is based on previous studies that have used bicarbonate infusion in the context of rhabdomyolysis secondary to compartment syndrome, finding a lower incidence of renal failure. Due to the aforementioned, we propose to carry out a similar intervention at the General Hospital of Mexicali, where there is a significant incidence of heatstroke during the summer months. The aim is to determine whether this intervention is useful in preventing the development of renal failure and the requirement for renal replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the General Hospital of Mexicali with the diagnosis of heat stroke.
* Meeting the operational definition (exposure to heat, body temperature at admission greater than 40 degrees Celsius).
* CPK level greater than 1000 U/L.
* Having informed consent from the patient or the legally responsible adult.

Exclusion Criteria:

* Exclusion of the heat stroke diagnosis during their evaluation.
* Lack of serum creatinine levels at the time of admission to the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
The use of sodium bicarbonate reduces the need for renal replacement therapy | From enrollment until discharge or death.
  Determine if the use of sodium bicarbonate as a prophylactic measure reduces the need for renal replacement therapy in patients with heat stroke-associated rhabdomyolysis.

SECONDARY OUTCOMES:
Creatinine levels | From enrollment until discharge or death.
  Describe the creatinine levels of patients diagnosed with heat stroke at the General Hospital of Mexicali.
Mortality rate | From enrollment until discharge or death.
  Determine the mortality rate of patients admitted with the diagnosis of heat stroke at the General Hospital of Mexicali.
Mortality rate of patients diagnosed with heat stroke who were administered bicarbonate compared to those who did not receive bicarbonate. | From enrollment until discharge or death.
  Determine the mortality rate of patients diagnosed with heat stroke who were administered bicarbonate compared to those who did not receive bicarbonate.
Potassium levels in patients diagnosed with heat stroke who received bicarbonate compared to those who did not receive bicarbonate. | From enrollment until discharge or death.
  Describe the potassium levels in patients diagnosed with heat stroke who received bicarbonate compared to those who did not receive bicarbonate.
Difference in the length of hospital stay for patients diagnosed with heat stroke who received bicarbonate compared to those who did not receive bicarbonate. | From enrollment until discharge or death.
  Determine if there is a difference in the length of hospital stay for patients diagnosed with heat stroke who received bicarbonate compared to those who did not receive bicarbonate.
Difference in the requirements for vasopressors in patients diagnosed with heat stroke who received bicarbonate compared to those who did not receive bicarbonate. | From enrollment until discharge or death.
  Establish if there is a difference in the requirements for vasopressors in patients
Use of mechanical ventilation in patients diagnosed with heat stroke | From enrollment until discharge or death.
  Establish if there is a difference in the use of mechanical ventilation in patients diagnosed with heat stroke who received bicarbonate compared to those who did not receive bicarbonate.

CONTACTS AND LOCATIONS:
Overall Officials: Hiram J Jaramillo Ramirez, MD, Principal Investigator — Hospital General de Mexicali
Locations (1):
- Hospital General de Mexicali, Mexicali, Estado de Baja California, Mexico

IPD SHARING:
Plan to Share IPD: No
There will be no disclousure of the patients information to thrid party members.

REFERENCES:
- [Background] Bouchama A, Knochel JP. Heat stroke. N Engl J Med. 2002 Jun 20;346(25):1978-88. doi: 10.1056/NEJMra011089. No abstract available. PMID 12075060